CLINICAL TRIAL: NCT05948735
Title: Construction and Assessment of an Intervention Model for Preventing Falls in Older Adults That Integrates Physiotherapy Exercise and Dance Movement Therapy
Brief Title: An Intervention Integrating Physical Therapy Exercise and Dance Movement Therapy for Preventing Falls in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Michal Elboim, Ph.D. - Physical Therapy Department, Faculty of Social Welfare & Health Sciences, University of Haifa, Haifa, Israel, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHaifa ME-G ESE MPB
Record Dates: First submitted 2023-06-19; First posted 2023-07-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2023-07

CONDITIONS: Older Adults
Keywords: Older adults; Fall; Fall prevention intervention; Physical therapy; Dance movement therapy; Otago Exercise Program
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the allocation to groups, and investigator will not be involved in the intervention process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Therapy Exercise and Dance Movement Therapy (PTE+DMT) (Experimental): The intervention include 12 face-to-face group sessions of 45 minutes each, twice a week for 6 weeks. The intervention integrates Otago Exercise Program (OEP)-based techniques and DMT techniques to address the emotional experience that arises during physical exercise. This include encouragement for spontaneous and creative movement on the part of the participants, and an invitation to verbally share the feelings, sensations, and thoughts that arose in the participants following the movement. At the end of the sessions, participants will be instructed to perform nine exercises independently at home, at a minimum of twice per week for six months
  Interventions: Other: Physical Therapy Exercise and Dance Movement Therapy (PTE+DMT) for Preventing Falls
- Physical Therapy Exercise (PTE) (Active Comparator): The intervention include 12 face-to-face group sessions of 45 minutes each, twice a week for 6 weeks. The intervention include OEP-based techniques only. At the end of the sessions, participants will be instructed to perform nine exercises independently at home, at a minimum of twice per week for six months.
  Interventions: Other: Physical Therapy Exercise (PTE) only for Preventing Falls

INTERVENTIONS:
Other: Physical Therapy Exercise and Dance Movement Therapy (PTE+DMT) for Preventing Falls — The intervention include 12 face-to-face group sessions of 45 minutes each, twice a week for 6 weeks. The intervention integrates OEP-based techniques and DMT techniques to address the emotional experience that arises during physical exercise. This include encouragement for spontaneous and creative movement on the part of the participants, and an invitation to verbally share the feelings, sensations, and thoughts that arose in the participants following the movement. At the end of the sessions, participants will be instructed to perform nine exercises independently at home, at a minimum of twice per week for six months.
  Arms: Physical Therapy Exercise and Dance Movement Therapy (PTE+DMT)
Other: Physical Therapy Exercise (PTE) only for Preventing Falls — The intervention include 12 face-to-face group sessions of 45 minutes each, twice a week for 6 weeks. The intervention include OEP-based techniques only. At the end of the sessions, participants will be instructed to perform nine exercises independently at home, at a minimum of twice per week for six months.
  Arms: Physical Therapy Exercise (PTE)

SUMMARY:
The goal of this study is to construct and assess a theoretical and interventional model for preventing falls in older adults that integrates physiotherapy exercise and dance movement therapy.

The main questions this study aims to answer are:

1. What is the effect on reducing fall risk in older adults of a group intervention focused solely on physical exercises, compared to a similar intervention that incorporates emotional content through dance movement therapy?
2. What are the factors of change in an intervention that integrates physical exercises and emotional content?
3. Is there a correlation between the outcome variables and the process variables in the study?

Researchers will compare: (1) an intervention group that integrates physical therapy exercises (PTE) and dance movement therapy (DMT), and (2) a PTE control group, to examine the effects on: (1) physical, (2) emotional, and (3) adherence to treatment.

DETAILED DESCRIPTION:
First, an invitation to participate in the study will be published through day centers and associations for older adults. Any participant who expresses interest in participating will receive a phone call from a researcher who is not involved in the intervention. During the call, they will receive a detailed explanation of the study. Additionally, an initial screening test will be conducted to determine the inclusion and exclusion criteria. Participants who meet the criteria will be asked to obtain permission from their family doctor to participate in group physical activity sessions aimed at preventing falls.

Second, each participant will be required to sign an informed consent form and complete a socio-demographic characteristics questionnaire during a meeting with the research coordinator held at the participants' day centers. Subsequently, a research assistant, who is not involved in the intervention, will conduct pre-intervention tests at the day centers. These tests will last approximately an hour and will involve administering questionnaires related to fall risk, daily functioning, fear of falling, falls-efficacy, perception of health status, depression, and the participants' expectations of the intervention. If needed, the research assistant will assist participants in reading and marking their answers to ensure consistency in how the questions are presented, taking into account each participant's level of attentiveness.

In addition, a research assistant with a bachelor's degree in physical therapy will perform two objective measurements to assess the participants' balance level using the Timed Up and Go (TUG) test and the Five Times Sit to Stand (5STS) test. Following the tests, the participants will be randomly assigned to groups using a random number table.

Each intervention group will consist of eight participants to allow the facilitator to address all participants and ensure their safety. The participants will attend 12 face-to-face group sessions, meeting twice a week for 6 weeks. The sessions will take place in suitable-sized rooms in the day centers visited by the participants. After each session, the group facilitator will complete a questionnaire to assess the adherence to the protocol (treatment fidelity), which will be reviewed by supervisors. Additionally, at the end of the second and fourth weeks, a research assistant will conduct a mid-test via telephone with the intervention groups participants, focusing on their experience of the treatment, satisfaction with the intervention, the therapist-patient relationship, and open-ended questions to evaluate the nature of the intervention.

At the end of the intervention, all groups will be instructed to independently perform the structured home practice exercises twice a week for the next six months, starting one week after the end of the intervention.

Within a week after the intervention concludes, each participant will undergo the same series of tests conducted prior to the intervention by the same research assistants. Furthermore, process indicators will be assessed. A telephone follow-up will be conducted once a week for a month by the research assistant to evaluate the participants' adherence to the home practice program. This follow-up will involve a structured questionnaire assessing the number of practice days per week and the number of exercises performed. At the end of the month, an open-ended question will be asked to evaluate the quality of the intervention for the intervention group participants. One month, two months, and six months after the intervention concludes, the research assistant will administer the questionnaires related to fear of falling, falls-efficacy, depression, and adherence to home physical activity via telephone to all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling adults aged 65 years or older.
2. Ability to independently walk for at least 10 meters with or without an assistive device.
3. Ability to walk for 2 minutes without an assistive device.

Exclusion Criteria:

1. Heart disease or respiratory disease.
2. A history of stroke, Parkinson's, or any other neurological disorder affecting walking.
3. Blindness or deafness that would prevent safe walking and hearing instructions.
4. A vestibular disorder such as vertigo.
5. Acute joint or musculoskeletal pain in the lower limbs that would limit continuous walking for 2 minutes.
6. Significant sensory problems in the lower limbs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Fall Risk Self-Assessment from baseline at 6 weeks | Pre- and post-intervention: within 5 days before the intervention (baseline), and within 5 days after the intervention (after 6 weeks).
  Fall risk assessment will perform using the Fall Risk Self-Assessment Tool (FRQ), which is a self-report questionnaire that includes 12 items rated on a dichotomous scale of "yes" or "no". The overall score of the questionnaire is the sum of the items to which the answer is "yes", and the score range is between 0 and 14. A score of 4 or higher indicates a level of risk of falling that requires a visit to a healthcare provider.
Change in Functional Status Questionnaire - Basic Activities of Daily Living (ADL) from baseline at 6 weeks | Pre- and post-intervention: within 5 days before the intervention (baseline), and within 5 days after the intervention (after 6 weeks).
  An assessment of Functioning in ADL will perform using the Functional Status Questionnaire-Basic ADL, which is a self-report questionnaire, specifically the functional assessment of performing activities in daily life (Activities of Daily Living [ADL]). The questionnaire includes a "Basis ADL" subscale, which consists of three items rated on a 5-point ordinal scale ranging from 0 (mostly did not perform due to other reasons) to 4 (mostly without difficulties), reflecting the degree of difficulty the individual experiences in performing daily activities such as eating, dressing, and bathing. The general score of the questionnaire scale was calculated by ((sum of items/number of items) - number of items) * (100/number of items), yielding a score range of 0 to 100, with a higher score indicating higher functional capacity. A score range between 0 and 87 is considered a warning zone and indicates a possibility of danger.
Change in Timed Up and Go test from baseline at 6 weeks | Pre- and post-intervention: within 5 days before the intervention (baseline), and within 5 days after the intervention (after 6 weeks).
  Objective balance assessment will perform using the Timed Up and Go (TUG) test. The time taken by participants while rising from a chair (46 cm height), for walking 3 m, turning, walking back, and sitting down, was measured. The TUG is conducted twice, and the average of the two test scores determine the overall score. A score higher than 13.5 seconds indicates a risk of falling among community-dwelling older adults
Change in Five Times Sit to Stand (5STS) test from baseline at 6 weeks | Pre- and post-intervention: within 5 days before the intervention (baseline), and within 5 days after the intervention (after 6 weeks).
  Objective balance assessment will perform using the Five Times Sit to Stand (5STS) test. The time taken by participants while getting up from a seated position in a chair and standing up and sitting down five times, was measured. Norm scores for ages 70 to 79 and 80 to 89 are 12.6 seconds and 14.8 seconds, respectively.
Change in Fear of Falling single item question from baseline at 6 months | Pre- and post-intervention: within 5 days before the intervention (baseline), and within 5 days after the intervention (after 6 weeks). Also, one month, two months, and six months after the intervention.
  Fear of Falling assessment will perform using the FOF single item question (FOF SIQ) which is a single self-report question: "Are you afraid of falling?". The question is rated on a Likert-type scale ranging from 1 (no, not afraid) to 4 (yes, indeed afraid).
Change in Short Falls Efficacy Scale-International from baseline at 6 months | Pre- and post-intervention: within 5 days before the intervention (baseline), and within 5 days after the intervention (after 6 weeks). Also, one month, two months, and six months after the intervention.
  Falls Efficacy assessment will perform using the Short Falls Efficacy Scale-International (Short FES-I), which is a self-report questionnaire that includes seven items rated on a Likert-type scale ranging from 1 (not at all concerned) to 4 (extremely concerned). The overall score of the questionnaire is the sum of its items, and the score range is be-tween 7 and 28. A lower score indicates better self-efficacy related to falls.
Change in The Patient Health Questionnaire from baseline at 6 months | Pre- and post-intervention: within 5 days before the intervention (baseline), and within 5 days after the intervention (after 6 weeks). Also, one month, two months, and six months after the intervention.
  Depression Assessment Questionnaire assessment will perform using the Patient Health Questionnaire (PHQ-9), which is a self-report questionnaire used to assess the presence and severity of depression. It consists of 9 items that list major depressive symptoms, based on the Diagnostic and Statistical Manual of Mental Disorders, and are rated on a 4-point scale ranging from 0 (not at all) to 3 (almost every day). The overall score of the questionnaire is calculated by summing the scores of all items and ranges from 0 to 27, with a higher score indicating a higher level of distress and depression. The researchers propose the following levels of depression: score 0 to 5 indicates absence of depression; score 6 to 9 indicates subsymptomatic/low depression; score 10 to 14 indicates moderate depression; score 15 to 19 indicates moderate-severe depression; and score 20 to 27 indicates severe depression.
Change in 12-item Short Form Health Survey (SF-12) from baseline at 6 weeks | Pre- and post-intervention: within 5 days before the intervention (baseline), and within 5 days after the intervention (after 6 weeks).
  Self-perceived health status assessment will perform using the 12-item Short Form Health Survey (SF-12), which is a self-report questionnaire that includes 12 items that are summarized as two scores: the Physical Component Summary (PCS-12), which refers to the physical aspect of health status, and the Mental Component Summary (MCS-12), which refers to the mental aspect of health status. Four items are rated on a dichotomous yes/no scale, while the remaining items are rated on a Likert-type scale with response options ranging from 3 to 6. The average score in each component is 50, and the standard deviation is 10. The overall scores range from 0 to 100. A higher score indicates a better perception of health status and quality of life.
Change in Exercise Adherence Rating Scale (EARS) from 7 weeks after the intervention at 6 months | Post-intervention: once a week after the intervention. Also, one month, two months, and six months after the intervention.
  Weekly telephone follow-up will be conducted for a month after the end of the intervention to assess persistence in the home practice program, including the number of days of practice per week and the number of exercises performed. In addition, home exercise adherence assessment will performed using the Exercise Adherence Rating Scale (EARS), which assesses an individual's adherence to performing exercises which were instructed by healthcare professional to perform at home. This self-report questionnaire includes six items rated on a Likert-type scale ranging from 0 (Completely agree) to 4 (Completely disagree). In one item, the phrase "my healthcare professional" was replaced with "the group instructor" to align with the study. The overall score of the questionnaire is the sum of its items, and the score range is between 0 and 24. A higher score indicating a higher level of adherence to performing exercises at home.

SECONDARY OUTCOMES:
Therapeutic Bond | Mid-test and post-intervention: During Cycle 1 (each cycle is 42 days), on the 14th day, 28th day, and at the end of Cycle 1 on the 42nd day.
  Therapist-patient bond assessment will be performed using the Therapeutic Bond subscale of the 36-item Working Alliance Inventory. The therapeutic bond sub-scale is a self-report questionnaire that includes 12 items rated by the patient on a Lik-ert-type scale ranging from 1 (does not describe my feeling at all) to 5 (very much describes my feeling). The overall score of the questionnaire is the items average, and the score range is between 1 and 5. A higher score represents a stronger bond with the therapist.
Subjective Vitality Scale (SVS) | Mid-test and post-intervention: During Cycle 1 (each cycle is 42 days), on the 14th day, 28th day, and at the end of Cycle 1 on the 42nd day.
  The SVS is a self-report questionnaire used to assess subjective feelings of aliveness during the intervention sessions. It consists of 7 items rated on a Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree) in reference to the participant's feelings during the sessions. The overall score of the questionnaire is calculated as the average of all items, and the score range is from 1 to 7, where a higher score indicates a higher level of perceived vitality.
Patient's Expectations | Pre-intervention, mid-test, and post-intervention:Before Cycle 1 (each cycle is 42 days), during Cycle 1 on the 14th day, 28th day, and at the end of Cycle 1 on the 42nd day.
  A self-report question to assess the patient's expectations from the intervention will be administered prior to the start of the intervention program (pre-test). The question is: 'To what extent do you believe that the sessions will help you feel better?' The response options are rated on a 3-point scale: 1 (not at all), 2 (to a moderate extent), or 3 (to a very large extent). weekly during the intervention period (mid-test), and after completing the intervention program (post-test), the patient will rate whether the intervention met their expectations on a 3-point scale: 1 (lower than expected), 2 (as expected), or 3 (higher than expected).
Assessment of the quality of the intervention | Mid-test and post-intervention: During Cycle 1 (each cycle is 42 days), on the 14th day, 28th day, and at the end of Cycle 1 on the 42nd day.
  Participants will undergo an open questions, telephone-based to evaluate their personal experience during the intervention period and afterwards, as part of an assessment of the quality of the intervention program. During the intervention period, participants will be asked two questions: "What was meaningful to you in the sessions this week?" and "What was significant to you in guiding the sessions this week?". After the intervention period, participants will be asked three questions: "What was most meaningful to you in the sessions?", "How did the sessions affect you physically?" and "How did the sessions affect you emotionally?". Additionally, one month after the end of the intervention, each participant will be asked: "What do you remember most from the meetings? And why?".

CONTACTS AND LOCATIONS:
Overall Officials: Michal Pitluk Barash, Principal Investigator — Faculty of Social Welfare & Health Sciences, University of Haifa
Locations (1):
- "Shalhevet" and "Savion" day centers; "Milav" social clubs, Kiryat Tivon; Yokneam; Haifa, Israel

IPD SHARING:
Plan to Share IPD: No